CLINICAL TRIAL: NCT04223089
Title: Accuracy of Transcutaneous Oxygen Monitoring (TCOM) vs Near Infrared Spectroscopy (NIRS) in Predicting Wound Outcomes in Patients Treated With or Without Revascularization
Brief Title: Accuracy of TCOM vs NIRS in Predicting Wound Outcomes in Patients Treated With or Without Revascularization
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00144156
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Wound Heal
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Revascularization: This group will include patients whose cutaneous oxygen partial pressure (PO2) around the wound of interest measures less than 40 mmHg and therefore require revascularization.
  Interventions: Diagnostic Test: Near Infrared Spectroscopy
- Medical Management: This group will include patients whose cutaneous PO2 around the wound of interest measures greater than 40 mmHg and will be managed conservatively in wound clinic
  Interventions: Diagnostic Test: Near Infrared Spectroscopy

INTERVENTIONS:
Diagnostic Test: Near Infrared Spectroscopy — The Kent Camera is intended for use by healthcare professionals as a non-invasive tissue oxygenation measurement system that reports an approximate value of the following in superficial tissue:
  * oxygen saturation (StO2),
  * relative oxyhemoglobin level (HbO2), and
  * relative deoxyhemoglobin (Hb) level
  The Kent Camera displays two-dimensional color-coded images of tissue oxygenation of the scanned surface and reports multispectral tissue oxygenation measurements for selected tissue regions. The Kent Camera is indicated for use to determine oxygenation levels in superficial tissues.

SUMMARY:
The primary purpose of this project is to compare the accuracy of transcutaneous oxygen monitoring and near infrared spectroscopy in assessing cutaneous oxygen levels in chronic wounds of patients following revascularization procedures as well as those with conservatively managed chronic wounds. This study will also compare the efficiency and practicality of both methods in guiding treatment decisions and management of these wounds.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18-85
* Presented with a non-healing lower extremity wound and have a Wagner classification for wound healing of grade 1 or 2

Exclusion Criteria:

* Wagner grade 3-5
* Congestive heart failure (CHF) with a left ventrical ejection fraction (LVEF) < 30%
* Have had a below the knee drug eluting stent placed (paclitaxel is chemo, can make wounds worse)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will include up to 200 adult patients who present with non-healing lower extremity wounds to the University of Kansas Medical Center. Patients will be grouped into two study arms depending on the degree of tissue ischemia (above or below 40 mmHg) and required treatment (conservative wound care alone or revascularization). Relevant clinical information will be obtained from patients' medical records including demographics, clinical history, intervention details, surgical records, and imaging data. Wound healing will be assessed at presentation, at the time of revascularization (pre and post-operative), and every 6 weeks thereafter by clinical assessment, Wagner classification, TCOM PO2 measurements and NIRS PO2 measurements. TCOM will guide treatment decisions and management, which is the current standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of NIRS measurements | From presentation to wound healing or amputation (approximately 6 months at most)
  To determine the accuracy of near infrared spectroscopy when compared to transcutaneous oxygen monitoring in assessing cutaneous oxygen levels and guiding treatment in patients with revascularized tissues or conservatively managed chronic wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Alli, MD, Principal Investigator — KUMC
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No